CLINICAL TRIAL: NCT05642715
Title: Trial of a Harm Reduction Strategy for People With HIV Who Smoke Cigarettes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Westat (Other); Massachusetts General Hospital (Other); Truth Initiative (Other); National Cancer Institute (NCI) (NIH); Red Planet Testing (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-14572; R01CA275521 (NIH)
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Hiv; Tobacco Use
Keywords: HIV; Tobacco; Cigarette; Smoking; Harm reduction
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tobacco Use; Smoking; Harm Reduction | interventions — Varenicline; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The treatment allocation will be concealed from the individual completing study assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EX+/HR (Experimental): The harm reduction arm (described in detail elsewhere)
  Interventions: Behavioral: EX+; Drug: Varenicline; Behavioral: HR
- EX+/TAU (Active Comparator): The treatment as usual arm
  Interventions: Behavioral: EX+; Drug: Varenicline; Behavioral: TAU

INTERVENTIONS:
Behavioral: EX+ — All participants, regardless of study arm, will be offered: BecomeAnEX, an online tobacco treatment with support community PLUS Positively Smoke Free on the Web (an intervention targeting people with HIV who smoke) integrated into the BecomeAnEX site.
  Other Names: BecomeAnEX+
Drug: Varenicline — All participants, regardless of study arm, will be offered: A 12-week course of varenicline dosed according to product label.
Behavioral: HR — Participants allocated to the EX+/HR arm will be offered: 30-minute video urging smokers who cannot or will not quit to cut down on cigarettes, and also to control their risk for lung cancer and cardio or cerebrovascular disease by undergoing low-dose CT screening for lung cancer (for those meeting prespecified criteria), and referral to Cardiometabolic Clinic (for those meeting prespecified criteria).
  Other Names: Harm Reduction
  Arms: EX+/HR
Behavioral: TAU — Participants allocated to the EX+/TAU arm will be offered: Medical treatment as usual from their regular providers after completing Stage 1 of the study
  Other Names: Treatment As Usual
  Arms: EX+/TAU

SUMMARY:
Cigarette smoking is now the leading killer of people with HIV (PWH) in the US, and most cessation strategies tried to date have failed to increase long-term quit rates. An "all or none" approach to smoking cessation in PWH offers little benefit to the large majority of PWH who are unable or unwilling to quit. In this proposal we argue that a harm reduction approach (i.e., cut down, get screened for lung cancer, control your blood pressure and cholesterol) has the potential to yield significant benefits in terms of the private and public health of PWH in the US.

DETAILED DESCRIPTION:
This will be a single-center, prospective, randomized controlled trial (RCT) enrolling 400 participants who are living with HIV and smoke cigarettes in the Bronx, New York. The vast majority (~85%) of people with HIV (PWH) who smoke and receive intensive cessation treatment combining behavioral and drug treatment (such as varenicline or nicotine patches) continue to smoke. The overall goal of this RCT is to compare a harm reduction (HR) strategy aimed at mitigating the harms of cigarette smoking, such as lung cancer and heart disease, in all PWH smokers, both those who are able to quit and those who continue smoking versus treatment as usual (TAU). All participants will have their blood pressure (BP) and lipid (cholesterol) profile checked at baseline. All participants will complete a questionnaire about their sociodemographic, clinical, and tobacco behavior histories at baseline, 3-months, 6-months, and 9-months. All participants who enroll in the trial will be randomized 1:1 (like a coin-flip) to the HR arm, called EX+/HR in this proposal, or the TAU arm, called EX+/TAU in this proposal. All participants will be offered intensive cessation treatment immediately after enrollment in the form of the BecomeAnEX+ online tobacco treatment program, which includes the web's largest online support community of people trying to quit, and an offer of a 12-week supply of varenicline. This stage of the trial, Stage 1, will extend from enrollment until 90-day post-enrollment. After that, in Stage 2, participants will be informed of their randomization assignment, i.e. to EX+/HR or EX+/TAU. Those who are assigned to EX+/HR will undergo the following: (A patient navigator [PN] will be assigned to each EX+/HR participant in order to facilitate all of the following activities.)

1. Harm reduction (HR) counseling. A 30-minute videosession that will emphasize abstinence as the best outcome, and that those who have quit should strive to remain abstinent for life. For those who have not quit, and mindful of the frequency of relapse in those who have, the video will provide rationale for cutting down, will detail the likely benefits associated with reduction in order to increase motivation, and will suggest specific strategies that are commonly employed in reduction interventions, namely (1) choosing specific cigarettes during the day to give up (2) increasing time intervals between cigarettes (3) smoking only during even or odd hours (4) restricting smoking to certain places (5) delaying the first cigarette of the day and (6) trying to avoid smoking completely on certain days. The video will go on to explain the importance of lung cancer screening and BP and lipid control in both selected smokers and ex-smokers and review the resources available to accomplish these goals, i.e. LDCT screening, Cardiometabolic (CM) Clinic, and patient navigator (PN) services.
2. Evaluation of eligibility for LDCT screening and referral for those who meet eligibility criteria. These criteria, based upon expert opinion and population-based modeling, will be age≥45 years and history of ≥20 pack years of smoking. From the investigators' pilot data the investigators expect 30.1% of enrollees to be ≥45 years old AND have a ≥20 pack year smoking history, and only 6.6% of these LDCT-eligible individuals will be 45-49 years of age. The project will conservatively budget for 10 scans to be paid for from research funds since individuals who meet CMS criteria for lung cancer screening (i.e. age ≥50 and ≥20 pack years smoking history) will have their scans paid for by their own medical insurance. The PN will schedule a LDCT, make reminder calls, ensure that transportation to the study is available (the study will provide fare cards) for these individuals, and inform their primary care providers of scan results. Although the investigators expect few, if any, referrals to originate from the EX+/TAU group, the study staff will log these events, and radiology staff will be blinded to study condition.
3. Evaluation of BP and cholesterol measurements and referral of individuals with SBP>130mmHg and/or LDL cholesterol>100mg/dl to CM Clinic, which provides expert management of these conditions. Based upon pilot data, the investigators expect 45.8% and 50.6% of the study cohort to have SBP>130mmHg and/or LDL>100mg/dl respectively. The investigators selected these BP and LDL cutoffs because it is unlikely that the specialty clinic will prescribe or modify any specific HTN or lipid treatment for measures below these values.

Cardiometabolic (CM) Clinic meets every Friday in the MMC outpatient department, and the PN will, similarly, arrange these appointments. Its mission is to optimize the CM profiles of its patients. This includes BP and lipid control. It is supervised by senior cardiology staff but also employs the services of specialized nursing, a dietitian, and an endocrinologist. Initiation and/or adjustment of antihypertensive medications and lipid management occurs directly in the clinic, with a note sent through the electronic health record (EHR) to the primary care provider. A single episode of brief cessation counseling is done for current smokers. Referrals for additional testing, such as ambulatory BP monitoring are made by the CM Clinic staff. Although the investigators expect few, if any, referrals to originate from the EX+/TAU group, study will log these events, and the clinic staff will be blinded and will not be informed which referred patients are participating in the trial.

Those who are assigned to the EX+/TAU group will undergo the following:

Participants allocated to EX+/TAU will continue to receive care from their primary care providers (PCP). A hard copy of the baseline and follow-up BP and lipid measurements will be delivered to the PCPs. Those who meet CMS criteria for LDCT screening and do not undergo screening during the trial will be offered a referral after their final study visit (these individuals will be eligible to undergo LDCT screening during their participation in the trial if they are referred by their care providers). LDCT screening and CM Clinic referral are fully available in ID Clinic, but they are barely utilized. In the first 6 months of 2021, only one clinic patient, out of more than 3000, completed LDCT screening, and only one clinic patient completed a visit to CM Clinic. As a result, even though LDCT screening and CM Clinic are available to ID Clinic patients, we expect to have good separation between study arms for comparison. The main outcomes to be compared between the two groups are summarized in the Outcome Measures module.

One of the great strengths of this trial is the investigators' partnership with the Cost-Effectiveness of Preventing AIDS Complications (CEPAC) group at the Massachusetts General Hospital. The CEPAC group is a national leader in modeling cost-effectiveness and health impact of treatment strategies for PWH to estimate their effects if deployed on a national level. The investigators will share the cost and outcome data that is accumulated in the course of the trial in order to enable sophisticated cost-effectiveness modeling. If, as the investigators expect, the HR approach is shown to be cost-effective, the modeling algorithms are equipped to estimate the potential number of lung cancer and cardiovascular deaths averted and years of life saved.

Finally, the investigators will employ the RE-AIM (reach, effectiveness, adoption, implementation, maintenance) framework to conduct a rigorous assessment of the practicalities and challenges associated with adopting an HR approach within a clinical setting.

Following an amendment approved by the IRB on 8/7/2025, recruitment efforts will be expanded as follows: a list of patients within the Montefiore Health System HIV Clinical Cohort Database who are classified as current smokers will be obtained through a query of the database conducted by the Einstein Epidemiology Informatics Study Management Unit (EISMU). These individuals will be contacted by telephone and/or mail to inform them of the trial and to offer them the opportunity to undergo screening and enrollment (if eligible).

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-79 (the ACC/AHA PCEs risk score is only valid in this age range).
2. Current cigarette smoking ("Yes" to: "Have you smoked more than 100 cigarettes in your lifetime?" AND "Have you smoked a cigarette, even a puff, in the past 7 days?" and have exhaled carbon monoxide (ECO) level ≥ 6ppm
3. Lab-confirmed HIV infection
4. Willingness to participate in a web-based tobacco treatment (EX+) AND offer of varenicline
5. Access to internet at least weekly and ability to read at ≥7th grade level (necessary to participate fully in EX+ program).
6. Willingness to be randomized to one of the two study conditions

Exclusion Criteria:

1. Pregnancy
2. Lack of insurance for specialty referral (we expect this exclusion to be rare because the great majority of people with HIV (PWH) at the Montefiore Medical Center have Medicaid or AIDS Drug Assistance Program (ADAP)
3. Contraindication to varenicline
4. Concurrent receipt of other cessation treatments
5. Evaluation in Cardiometabolic Clinic within the 12 months prior to enrollment
6. To minimize study contamination, eligible individuals who are spouses, partners, or roommates of participants will be excluded

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in cigarettes smoked per day (CPD) | From baseline to 9 months
  Change in the number of cigarettes smoked per day (CPD) from baseline will be determined. Results will be summarized by study arm using basic descriptive statistics. The study will have 80% power to detect a difference of 3.4 CPD between the two study conditions.
Occurrence of low-dose CT (LDCT) screening for lung cancer | Up to 9 months
  Occurrence of low-dose CT screening for lung cancer will be assessed by determining the number/percentage of participants who complete LDCT screening for lung cancer. Results will be summarized by study arm/group. The study will have 80% power to detect a difference in percentage completing screening between the two study conditions if ≥ 9.8% of the EX+/HR participants complete screening.
Change in systolic blood pressure (SBP) | From baseline to 9 months
  Change in systolic blood pressure (SBP) will be evaluated. All participants will have blood pressure checked at baseline, 6 months, and 9 months. Results will be summarized by study arm using basic descriptive statistics. The study will have 94.5% power to detect the expected difference of 7.7mmHg in SBP between the two study conditions.
Change in total cholesterol | From baseline to 9 months
  Change in total cholesterol from baseline will be evaluated. Blood samples will be collected as part of the lipid profile and samples will be submitted for laboratory analysis. Results will be summarized by study arm using basic descriptive statistics. The study will have 98.6% power to detect the expected difference of 21.5mg/dl in total cholesterol between the two study conditions.
Change in American College of Cardiology/American Heart Association Pooled Cohort Equation score (ACC/PCEs) | From baseline to 9 months
  Change in cardiovascular risk score from baseline will be determined based on American College of Cardiology/American Heart Association (ACC/AHA) Pooled Cohort Equation (PCE) score for risk of atherosclerotic cardiovascular disease (ASCVD). PCE score will be assessed at baseline, 6 months, and 9 months. The ACC/AHA PCEs are calculators used to estimate the 10-year risk of ASCVD (i.e., heart attack, stroke) for primary prevention, using factors like age, sex, race, cholesterol, blood pressure, diabetes, and smoking status. Results will be summarized by study arm using basic descriptive statistics. The study will have 80% power to detect a difference of 3.0 in PCEs score between the two study conditions.
Biochemically-confirmed 7-day point-prevalence abstinence (PPA) | 9 months
  Abstinence from tobacco smoking will be evaluated based on biochemically-confirmed 7 day PPA. Results will be summarized by study arm using basic descriptive statistics.

SECONDARY OUTCOMES:
Occurrence of Cardiometabolic Clinic appointment | 9 months
  Occurrence of Cardiometabolic Clinic appointment. Participants will be referred to Cardiometabolic (CM) Clinic for management of HTN [systolic BP>130mmHg] and/or hyperlipidemia [LDL cholesterol>100mg/dl]. Patient Navigators (PNs) will arrange for these appointments. The CM Clinic meets weekly in the MMC outpatient department. The number/percentage of participants who are referred to the CM clinic and attend their appointment will be summarized by study arm.
Proportion of participants at target systolic blood pressure | 9 months
  Proportion of participants achieving target systolic blood pressure will be evaluated. The target SBP is <=130mm/Hg. All participants will have blood pressure checked at 9 months. Results will be summarized by study arm using basic descriptive statistics.
Proportion of participants at target low dose low-density lipoprotein (LDL) cholesterol | 9 months
  Proportion of participants achieving target low dose low-density lipoprotein (LDL) cholesterol will be evaluated. The target LDL cholesterol is <=100mg/dl. Blood samples will be collected as part of the lipid profile at 9 months and samples will be submitted for laboratory analysis. Results will be summarized by study arm using basic descriptive statistics.
Change in CD4+ lymphocyte count | From baseline to 9 months
  Change in CD4+ lymphocyte count from baseline will be evaluated. Blood samples will be collected as part of the CD4+ count at 9 months and samples will be submitted for laboratory analysis. Results will be summarized by study arm using basic descriptive statistics.
Proportion with undetectable HIV-1 viral load | 9 months
  The proportion of participants with undetectable HIV-1 viral load at 9 months will be determined. Blood samples will be collected as part of the HIV-1 viral load at 9 months and samples will be submitted for laboratory analysis. Results will be summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shuter, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States